CLINICAL TRIAL: NCT02226432
Title: The Use of Antagonistic Muscle Magnetic Stimulation to Avoid Extensive Lesions and Improve Results of Selective Peripheral Neurotomy on Refractory and I POost Stroke Spasticity With Exclusive or Predominant Right Upper Limb Arm
Brief Title: Combined Antagonistic Muscle Magnetic Stimulation and Selective Periferal Neurotomy to Improve Results on Spasticity
Acronym: Andreani2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Juan Carlos M. Andreani MD (Other)
Responsible Party: Sponsor-Investigator, Juan Carlos M. Andreani MD, MD, Sociedad Argenttina de Neuromodulación
Organization: Sociedad Argenttina de Neuromodulación (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Andreani, JCM 2
Record Dates: First submitted 2014-08-16; First posted 2014-08-27 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: STROKE
Keywords: Barthel Scale; Disability; Modified Ashworth Scale; Right Arm; Neuromodulation; Spasticity; Stroke
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesics (Sham Comparator): - Classic Rehabilitation and Kinesic Therapy
  Interventions: Procedure: - Postoperative Antagonistic Peripheral Magnetic Stimulation; Other: Kinesics
- surgery (Sham Comparator): - Surgery:
  Selective Peripheral Neurotomy is surgical a method of section on suplying peripheral nerves of motor fascicles to relieve harmful spasticity. An intraoperative stimulation of motor fascicles is done, and those which abnormal spreading on far placed myotomes are more evident are chosen to be sectioned.
  Interventions: Procedure: - Postoperative Antagonistic Peripheral Magnetic Stimulation; Other: Kinesics
- Magnetic Stimulation (Active Comparator): - Postoperative Antagonistic Peripheral Magnetic Stimulation with 1.5 tesla intensity, infrathreshold 80 per cent of minimal intensity able to produce always muscle contraccion. Trials repeated twice a week in sessions of 30 minutes during 6 months
  Interventions: Procedure: - Postoperative Antagonistic Peripheral Magnetic Stimulation; Device: Selective Peripheral Magnetic Stimulation; Other: Kinesics

INTERVENTIONS:
Procedure: - Postoperative Antagonistic Peripheral Magnetic Stimulation — Selected patients will be treated with Selective peripheral Neurotomy followed by an standartized cycle of Selective Peripheral Magnetic Stimulation and classic post operative Kinesic Therapy.
  * Sham patients (n 10) will be treated with classic post operative Kinesic Therapy.
  * Comparision of both groups will be statistified
  Other Names: - Preoperative Peripheral Nerve Blockade; - Selective Peripheral Neurotomy; - Kinesic Rehabilitation Therapy
Device: Selective Peripheral Magnetic Stimulation — Peripheral 1.5 tesla intensity, 10 Hz of Frequency, with "eight saped" bovine, of 30 minutes, aplied on antagonistic muscles, twice a week. Intensity will be infrathreshold, 80 per cent of the individual threshold (minimal amount of intensity producing always a muscle motor response in each particular patient)
  Arms: Magnetic Stimulation
Other: Kinesics — Session of classic Kinetic Rehabilitation and motor exercises, twice a week on Physicians´s office and dayly on patient´s home.
  Other Names: Classic Rehabilitation Treatment

SUMMARY:
The objective of the present trial is to demonstrate Magnetic stimulation as an useful complementary treatment in order to improve patients' evolution without the need of extensive surgical lesion.

DETAILED DESCRIPTION:
Patients with refractory post stroke upper right limb spasticity will operated by Median nerve or Median/ Cubital selective neurotomy depending upon more affected territories.

Some of them could be also also operated with posterioris tibialis neurotomy to treat equine's foot whenever also clinically present. Preoperative motor blocks might be possitive in all cases.

A week later, they will be treated by magnetic stimulation on selected antagonistic muscles, related to pre - operative affected ones, mostly deltoids, triceps and finger extensors with an equipment Dipol Zeta D5 (Russian Federation), with 1.5 tesla of intensity.

Trials will be repeated twice a week in sessions of 30 minutes during 6 months with simultaneous intensive classic rehabilitation.

Patients will be monthly evaluated by the mean score of Modified Ashworth Scale, related to fingers, wrist, elbow and shoulder and also with Barthel Scale.

ELIGIBILITY:
Inclusion Criteria:

* Severe and refractory right Hemiparesia or Hemiplegia, affecting hand function.
* Failure of kinesic treatment
* 2 points or more Improvement on Modified Ashworth Scale after anestethic blockade

Exclusion Criteria:

* Severe cardiovascular disease
* Severe pulmonary disease
* Neoplasia advanced disease
* Joint anchylosis
* Irreversible retraction for muscle fibrosis

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | Post operative Modified Ashworth Scale /MAS) setted up monthly for each patient taking into account the postoperative date, during six continued months.
  - Mean Preoperative and sequencial monthly postoperative evaluation of stiffness and ranges of joint pasive movements at the shoulder, elbow, wrist and fingers.

SECONDARY OUTCOMES:
Fugl - Meyer Scale | Post operative Fugl - Meyer Scale evaluation, setted up monthly for each patient taking into account the postoperative date, during six continued months.
  Pre and post operative evaluation of a set of active and pasive movements and articular angles in the upper limb
Barthel Scale | Post operative Barthel Scale evaluation setted up monthly for each patient taking into account the postoperative date, during six continued months.
  Pre and post operative evaluation of ten basic current dayly life activities, scored 10, 5 or 0 points each one, a total of 100 points

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Mario Andreani, MD, Study Director — Fundación CENIT; Fabián César Piedimonte, MD, Principal Investigator — Fundación CENIT - President

IPD SHARING:
Plan to Share IPD: No